CLINICAL TRIAL: NCT02747654
Title: Development of a Dosing Model Based on Anti-tuberculosis Drug Monitoring NAT2 Genotypes in Tuberculosis Patients.
Brief Title: Isoniazid Dosage Prediction Model Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC-2013-07-155-002
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: NAT2 Genotype
Keywords: NAT2 genotype guided dosing
MeSH Terms: interventions — Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard dosing (No Intervention): a standard treatment group; INH dose of 300 mg or 200 mg based on the body weight
- Genotype-guided dosing (Experimental): INH dose determined based on developed model
  Interventions: Genetic: genotype

INTERVENTIONS:
Genetic: genotype — Patients were randomly assigned to a standard treatment group; INH dose of 300 mg or 200 mg based on the body weight) or model-based treatment group; INH dose determined based on developed model,
  Arms: Genotype-guided dosing

SUMMARY:
Isoniazid (INH) is an essential component of first-line anti-tuberculosis (TB) treatment. However, treatment with INH is complicated by polymorphisms in the expression of the enzyme system primarily responsible for its elimination, N-acetyltransferase 2 (NAT2), and its associated hepatotoxicity. The objective of this study was to develop an individualized INH dosing regimen using a pharmacogenetic-driven model and to apply this regimen in a pilot study.

ELIGIBILITY:
* Eligible participants were patients newly diagnosed with active TB
* Who underwent standard four drug treatment for 6months: isoniazid (5 mg/kg, usually 300 mg), rifampin (450 mg for <50 kg or 600 mg for 50 kg body weight), ethambutol(15mg/kg), and pyrazinamide (20 - 30 mg/kg)
* Given daily for two months and followed by isoniazid and rifampin with or without ethambutol for four months.
* Those patients with abnormal hepatic function on laboratory testing (increased serum aspartate aminotransferase, alanine aminotransferase, or total bilirubin) before anti-TB treatment, underlying liver disease or systemic illness such as congestive heart failure, acute life-threatening disease, or alcoholism, or disease that was resistant to INH at the start of treatment were excluded.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Serum concentrations of INH | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Youn Lee, MD, Principal Investigator — Sargodha Medical College
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No